CLINICAL TRIAL: NCT01756742
Title: Effectiveness of a Program of Respiratory Physiotherapy on Pleural Effusion: a Randomized Controlled Trial
Brief Title: Effects of Respiratory Physiotherapy on Pleural Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0038UG
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Pleural Effusion
Keywords: Pleural Effusion; Respiratory physiotherapy; Length of stay
MeSH Terms: conditions — Pleural Effusion | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Respiratory physiotherapy (Experimental): 54 people according to the inclusion criteria were recruited to have a respiratory physiotherapy treatment added to their medical intervention.
  Interventions: Other: Respiratory physiotherapy
- Conservative treatment (Placebo Comparator): 49 people were recruited in this group. These participants received conservative medical treatment intervention
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Other: Respiratory physiotherapy — The respiratory physiotherapy intervention included:
  * Mobilisation techniques: limb exercises (passive, active assisted, or active resisted)
  * Chest physiotherapy: it included a Controlled breathing program, pursed lips breathing (PLB), active expiration and incentive spirometry.
  Other Names: Respiratory techniques added to conservative treatment
  Arms: Respiratory physiotherapy
Other: Conservative treatment — Conservative medical treatment intervention for pleural effusion.
  Other Names: Medical treatment
  Arms: Conservative treatment

SUMMARY:
Pleural effusion and the complexity of diagnosis and treatment make planning and delivering care challenging. Respiratory physiotherapy is recommended, and should be applied during the first weeks of treatment.The aim of the present study is to demonstrate the effectiveness of a respiratory physiotherapy protocol in patients with Pleural Effusion who attended a University Hospital.

DETAILED DESCRIPTION:
Approximately 1.5 million patients are diagnosed with pleural effusion each year in the United States . Pleural effusion (PE) is an accumulation of fluid in the pleural space that is classified as transudate or exudate according to its composition and underlying pathophysiology. The goal in the management of pleural effusion is to provide symptomatic relief by removing fluid from the pleural space and to allow the treatment of the underlying disease. While some authors (REF) propose respiratory physiotherapy, in the majority of the cases only the medical treatment combined with the pleural fluid removal by thoracentesis are the most common practice. The objective of this study is verify the effectiveness of respiratory physiotherapy in pleural effusion

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pleural effusion based on the presence of a consistent radiological finding on simple posteroanterior and lateral chest X-rays, and decubitus lateral in cases of small PE.

Exclusion Criteria:

* Non diagnosis of pleural effusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the severity of respiratory disease | baseline, 12 months
  A spirometry is used to assess severity of individual patients respiratory disease and their response to therapy and is regarded as the gold standard measure of respiratory function. The following variables were recorded; forced vital capacity, forced expiratory volume achieved in 1 second, and the forced expiratory flow over the middle one half of the forced vital capacity.

SECONDARY OUTCOMES:
Length of the hospital stay | baseline, 12 months
  Length of stay was defined as the number of days between admission and discharge.
Severity in the pleural effusion repercussion | baseline, 12 months.
  The chest radiograph has been the initial diagnostic tool for the detection and evaluation of pleural effusion. The severity was codified from 0(normal) to 10 (very severe) by a radiologist with more than 8 years of experience.

CONTACTS AND LOCATIONS:
Overall Officials: M. Carmen Valenza, MD, Principal Investigator — Universidad de Granada
Locations (1):
- Universitary Hospital San Cecilio, Granada, Andalusia, Spain